CLINICAL TRIAL: NCT02476851
Title: Clinical Investigation to Evaluate the Haemonetics POLFA Modified Sample Needle Assembly With Vacuum Tube Holder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Haemonetics Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: TP-CLN-100380
Record Dates: First submitted 2015-06-11; First posted 2015-06-19 (Estimated); Results first posted 2022-04-29 (Actual); Last update posted 2022-04-29 (Actual); Status verified 2022-04

CONDITIONS: Transmission, Blood, Recipient/Donor
Keywords: Blood Donation; Whole Blood

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- POLFA (Experimental Needle Assembly) first, then Kawasumi (Control Needle Assembly) (Other): Ensure that whole blood passed through the POLFA needle assembly (the investigational needle assembly or "INA") has a supernatant hemoglobin within the acceptable range of < 100mg/dL. Each subject receives the same intervention (Standard of Care blood draw) and blood is drawn into both the INA and CNA. The difference is the order in which the CNA or INA is applied.
  Interventions: Device: POLFA (Needle Assembly); Device: Kawasumi (Needle Assembly)
- Kawasumi (Control Needle Assembly) first, then POLFA (Experimental Needle Assembly) (Other): Ensure that whole blood passed through the POLFA needle assembly (the investigational needle assembly or "INA") has a supernatant hemoglobin within the acceptable range of < 100mg/dL. Each subject receives the same intervention (Standard of Care blood draw) and blood is drawn into both the INA and CNA. The difference is the order in which the CNA or INA is applied.
  Interventions: Device: POLFA (Needle Assembly); Device: Kawasumi (Needle Assembly)

INTERVENTIONS:
Device: POLFA (Needle Assembly) — Each subject receives the same intervention and blood is drawn into both the INA and CNA. The difference is the order in which the CNA or INA is applied.
Device: Kawasumi (Needle Assembly) — Each subject receives the same intervention and blood is drawn into both the INA and CNA. The difference is the order in which the CNA or INA is applied.

SUMMARY:
This study evaluates whether whole blood transferred through the new POLFA needle assembly meets supernatant hemoglobin acceptability standards.

DETAILED DESCRIPTION:
The POLFA needle is part of the set's PPD (personal protection device) sampling port assembly that facilitates safer blood transfer between the collection set (i.e., the diversion pouch) and a Vacutainer® for the purpose of viral testing or other testing of the whole blood. The POLFA needle assembly was developed as a means to reduce costs while maintaining functionality, quality and safety. Since the overall functionality of the POLFA needle was designed to be equal to the currently approved Kawasumi needle, a change to the overall device safety and use profile is neither anticipated nor intended.

This trial will serve to generate data sufficient to demonstrate that blood transferred through the POLFA needle results in plasma hemoglobin levels below 100mg/dL.

ELIGIBILITY:
Eligibility Criteria:

* Study donor must be ≥ 18 years of age.
* Study donor must weigh ≥ 110 pounds.
* Study donor's body temperature must be ≤ 37.5°C / 99.5°F (oral).
* Study donor's hemoglobin must be ≥12.5 g/dL.
* Study donor's hematocrit must be ≥ 38%.
* Study donor must meet all criteria per respective site's Research Blood Donation Record (BDR).
* Study donor's most recent single RBC unit donation must have been ≥56 days prior to study donation.
* Study donor's most recent double RBC unit donation must have been ≥ 112 days prior to study donation.
* Study donor must have consented to study participation by reviewing and having expressed understanding the site-respective IRB-approved informed consent form prior to undergoing any study related procedures.
* Study donors must agree to report adverse events from the time of signing the informed consent to twenty-four hours following the end of their active study involvement.
* Study donors must not have experienced any of the following:

Physical trauma consistent with associated coagulopathy within the last 30 days, Surgery within the last 30 days, Known history of hypercoagulopathy (i.e., Factor V Leiden, Prothrombin G20210A, idiopathic venous thrombotic events, etc.).

* Female study donors must not be pregnant, expected to be pregnant or breastfeeding.

Exclusion Criteria - any individual not meeting the above criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2015-06; Primary Completion 2015-07 (Actual); Study Completion 2015-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lou Ann Maes, MD, Principal Investigator — American Red Cross Mid-Atlantic Region; Jose Cancelas, MD, Principal Investigator — Hoxworth Blood Center
Locations (3):
- United States (3):
  - Haemonetics, Braintree, Massachusetts
  - Hoxworth Blood Center, Cincinnati, Ohio
  - American Red Cross Mid-Atlantic Region Blood Services, Norfolk, Virginia

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | POLFA (Experimental Needle Assembly) First, Then Kawasumi (Control Needle Assembly) | Kawasumi (Control Needle Assembly) First, Then POLFA (Experimental Needle Assembly)
Started | 31 | 31
Completed | 30 | 30
Not Completed | 1 | 1
Not completed — Protocol Violation | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- POLFA (Experimental Needle Assembly) First, Then Kawasumi (Control Needle Assembly): Donors in this arm were randomized to have approximately half of their blood collection pass first through the POLFA Needle Assembly, and then through the Kawasumi Needle Assembly.
- Kawasumi (Control Needle Assembly) First, Then POLFA (Experimental Needle Assembly: Donors in this arm were randomized to have approximately half of their blood collection pass first through the Kawasumi Needle Assembly, and then through the POLFA Needle Assembly.
- Total: Total of all reporting groups
Arm/Group | POLFA (Experimental Needle Assembly) First, Then Kawasumi (Control Needle Assembly) | Kawasumi (Control Needle Assembly) First, Then POLFA (Experimental Needle Assembly | Total
Number analyzed (Participants) | 31 | 31 | 62
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.3 (13.4) | 47.1 (12.5) | 46.7 (12.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 15 | 34
  Male | 12 | 16 | 28
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 31 | 31 | 62
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 4 | 8
  White | 26 | 27 | 53
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 31 | 31 | 62
Body Temperature [Mean (Standard Deviation); unit: degrees F] | 98.0 (0.57) | 97.8 (0.55) | 97.9 (0.57)
Weight [Mean (Standard Deviation); unit: pounds] | 172.3 (33.5) | 186.4 (38.9) | 179.4 (36.7)
Height [Mean (Standard Deviation); unit: inches] | 66.2 (3.7) | 67.1 (3.5) | 66.7 (3.6)
Systolic Blood Pressure [Mean (Standard Deviation); unit: mmHg] | 128.4 (20.1) | 124.0 (17.8) | 126.2 (18.98)
Diastolic Blood Pressure [Mean (Standard Deviation); unit: mmHg] | 74.6 (10.5) | 73.3 (9.89) | 74.0 (10.1)
Pulse [Mean (Standard Deviation); unit: bpm] | 74.3 (10.3) | 74.7 (10.0) | 74.5 (10.1)
Donor Hemoglobin [Mean (Standard Deviation); unit: g/dL] | 14.2 (1.4) | 14.4 (1.1) | 14.3 (1.3)

OUTCOME MEASURES:

1. Primary Outcome: Plasma Supernatant Hemoglobin
Description: To determine whether whole blood transferred to a Vacutainer® through the POLFA needle will have supernatant hemoglobin levels <100 mg/dL within a 95% CI and 95% reliability. The average hemoglobin levels in the blood collected through each assembly is presented.
Time Frame: Following a one-time whole blood donation, samples were measured within 1 month of donation.
Population: Number of participants analyzed represents all participants that contributed blood to each assembly.
Measure: Mean (Standard Deviation); unit: mg/dL
Groups:
- POLFA (Experimental Needle Assembly): Blood was drawn through the experimental assembly and the hemoglobin levels were measured.
- Kawasumi (Control Needle Assembly): Blood was drawn through the control assembly and the hemoglobin levels were measured.
Arm/Group | POLFA (Experimental Needle Assembly) | Kawasumi (Control Needle Assembly)
Number analyzed (Participants) | 60 | 60
mg/dL | 26.8 (15.7) | 28.0 (14.6)

ADVERSE EVENTS:
Time Frame: Up to 24 hours following the end of study procedure (one-time whole blood donation).
Arm/Group | POLFA (Experimental Needle Assembly) | Kawasumi (Control Needle Assembly)
All-Cause Mortality (participants affected / at risk) | 0/60 | 0/60
Serious Adverse Events (participants affected / at risk) | 0/60 | 0/60
Other Adverse Events (participants affected / at risk) | 0/60 | 0/60

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No